CLINICAL TRIAL: NCT03680352
Title: Phase 1, Open-label, Parallel Group, Single-dose Study to Evaluate the Pharmacokinetics, Safety and Tolerability of AAI101 With Cefepime in Subjects With Varying Degrees of Renal Function
Brief Title: Pharmacokinetics of Cefepime and AAI101 in Subjects With Renal Insufficiency and Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Allecra (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: AT-102
Record Dates: First submitted 2018-07-25; First posted 2018-09-21 (Actual); Last update posted 2022-06-28 (Actual); Status verified 2022-06

CONDITIONS: PK in Patients With Various Degrees of Renal Impairment
MeSH Terms: interventions — Cefepime; enmetazobactam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- cefepime/AAI101 combination (Experimental): Investigational drug
  Interventions: Drug: cefepime/AAI101

INTERVENTIONS:
Drug: cefepime/AAI101 — Fixed dose combination of cefepime and AAI101

SUMMARY:
This is a Phase 1, multi-center, open-label, PK and safety study of a single dose of AAI101 in combination with cefepime in male and female subjects with mild renal impairment (Group 1, n = 6), moderate renal impairment (Group 2, n = 6), severe renal impairment (Group 3, n = 6), ESRD requiring dialysis (Group 4, n = 6), and normal renal function (Group 5, n = 6) as defined using the estimated value for creatinine clearance (CLcr) at Screening.

The study consists of a 28-day screening period, followed by a single dose administration of AAI101 in combination with cefepime antibiotic on Day 1, an in house period (assessment period) and follow-up visit. All subjects will be confined to the study site from Day -1 (the day before dosing) until the morning of Day 3. The follow-up visits will occur on Day 7 (±2 days), on Day 14 (±2 days), and on Day 30 (±2 days), if the results of the safety hepatic assessments are abnormal on Day 14 (±2 days).

Group 4 (ESRD requiring dialysis) will have 2 in-house periods (separated by at least 7 days), and will receive the single doses of AAI101 in combination with cefepime antibiotic once after dialysis and once before dialysis. The follow-up visit for Group 4 will occur on Day 7 (±2 days), on Day 14 (±2 days), and on Day 30 (±2 days), if the results of the safety hepatic assessments are abnormal on Day 14 (±2 days), counting from Day 1 of the second period.

ELIGIBILITY:
Main Inclusion Criteria

* Adult male or female subjects age 18 to 70 years, inclusive
* BMI 18.0 35.0 kg/m2, inclusive, where BMI (kg/m2) = body weight (kg) / height2 (m2) Subjects with Renal Impairment (in addition)
* Stable renal impairment, defined as no clinically significant change in disease status, as judged by the Investigator Healthy Subjects (in addition)
* Subjects with normal renal function as evidenced by CLcr
* Judged to be in good health in the opinion of the Investigator on the basis of a medical evaluation that reveals the absence of any clinically relevant abnormality OR Subject has a stable disease (e.g., hypertension, hyperlipidemia, diabetes mellitus, hyperthyreosis) under medical control.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
The maximum plasma concentration (Cmax) of cefepime and AAI101 | Up to 48 hours post-dose
  Cmax will be compared before and after administration of a single dose of cefepime/AAI101
AUC0-inf: area under the concentration-time curve (AUC) from time 0 extrapolated to infinity of cefepime and AAI101 | Up to 48 hours post-dose
  AUC0-inf will be compared before and after administration of a single dose of cefepime/AAI101

SECONDARY OUTCOMES:
The number of volunteers with adverse events as a measure of safety and tolerability | Up to 96 hours post-dose
  Assessments will be made via recording of AEs.

CONTACTS AND LOCATIONS:
Locations (2):
- Pharmaceutical Research Associates CZ, s.r.o., Prague, Jankovcova, Czechia
- PRA Magyarország Kft Fázis I-es Klinikai Farmakológiai Vizsgálóhely, Budapest, Rottenbiller Utca 13, Hungary

IPD SHARING:
Plan to Share IPD: No